CLINICAL TRIAL: NCT02671253
Title: Myomectomies:Tumor Characteristics and Clinical Implications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Päivi Päkarinen, MD PhD, Helsinki University Central Hospital
Other Study IDs: 24/13703/03/2015
Record Dates: First submitted 2016-01-25; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Uterine Myomectomy; Genetics; Quality of Life; Gynecologic Surgical Procedures
MeSH Terms: interventions — Uterine Myomectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Myomectomy — The patient series consists of consecutive patients scheduled for elective laparotomic, traditional laparoscopic or robotic assisted laparoscopic myomectomy. The surgical method is selected based on clinician´s preference.

SUMMARY:
This project focuses on myomectomy patients in reproductive age. The aim is to study both the molecular characteristics of uterine fibroids and to characterize the clinical effects of surgical treatment.

Patient series is mainly retrospective and consists of individuals who have undergone myomectomy at Helsinki University Central Hospital (HUCH) during 2009-2015. In addition, the investigators have started a prospective sample collection starting in October 2015, collecting samples from myomectomies.

Clinical data sources include medical records, specific questionnaires and a quality of life -questionnaire filled by patients.

ELIGIBILITY:
Inclusion Criteria:

* Uterine leiomyoma
* Seeking for surgery

Exclusion Criteria:

* Language proficiency in Finnish, Swedish or English

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women at age under 46 years undergoing myomectomy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life measured by a validated questionnaire (UFS-QOL) | Two years
  UFS-QOL: Uterine Fibroid Symptom and Health-Related Quality of Life Questionnaire

SECONDARY OUTCOMES:
Pregnancy rate after myomectomy, data collected with questionnaire | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Päivi I Pakarinen, MD PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Kätilöopisto Maternity Hospital, Helsinki University hospital, Helsinki, Huch, Finland

IPD SHARING:
Plan to Share IPD: No